CLINICAL TRIAL: NCT00002490
Title: A RANDOMIZED TRIAL OF RADICAL RADIOTHERAPY IN pT1G3 NXM0 BLADDER CANCER
Brief Title: Radiation Therapy, Chemotherapy, or Observation in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000077404; MRC-BS06; EU-91019; ISRCTN65282717
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2001-06

CONDITIONS: Bladder Cancer
Keywords: stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine; Mitomycin; Radiotherapy

INTERVENTIONS:
Biological: BCG vaccine
Drug: mitomycin C
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more tumor cells. It is not known whether receiving either radiation therapy, chemotherapy, or observation is more effective for cancer of the bladder.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy, chemotherapy, or observation following tumor surgery in treating patients who have bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of adjuvant radical radiotherapy vs intravesical BCG or mitomycin vs observation alone after endoscopic resection in terms of the progression rate and survival of patients with stage I, grade 3 transitional cell carcinoma of the bladder.
* Determine the toxicity of radical radiotherapy in these patients.
* Determine the incidence of carcinoma in situ elsewhere in the bladder and its correlation with the subsequent clinical outcome of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, extent of tumor (single tumor without carcinoma in situ (CIS) vs multiple tumors or CIS), and WHO performance status. Patients with a single tumor and no CIS are randomized to arm I or II. Patients with multiple tumors or CIS are randomized to arm II or III.

* Arm I: Patients undergo observation only.
* Arm II: Patients undergo radical radiotherapy 5 days a week for 6 weeks. Patients found to be node positive on CT scan may undergo pelvic irradiation and remain on study.
* Arm III: Patients receive intravesical BCG or mitomycin (at the discretion of the physician) weekly for 6-12 weeks.

Patients on arms I and III are followed at 3 months after randomization. All patients are followed at 6, 9, and 12 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of transitional cell carcinoma of the bladder

  * Stage T1 Nx M0, grade 3 disease
  * No muscle invasion at base of tumor
  * Diagnosis of this stage made within the past 6 months

    * Earlier diagnosis of tumors with lower stage or grade allowed
    * No history of higher stage urothelial tumors
* Presence of partial involvement of bladder with carcinoma in situ (CIS) or asymptomatic widespread CIS allowed

  * No widespread CIS causing severe symptoms
* Prior complete transurethral resection of tumor with deep biopsy of underlying bladder wall required
* Disease currently amenable to adjuvant radiotherapy, followed by cystoscopy with biopsies

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other prior or concurrent malignancy except nonmelanomatous skin cancer or cervical intraepithelial neoplasia

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 1 prior adjuvant treatment with intravesical BCG

Chemotherapy:

* No more than 1 prior adjuvant treatment with intravesical chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics
* Diathermic removal of associated small papillary growths allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-09

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Harland, MD, Study Chair — University College London Hospitals
Locations (1):
- Middlesex Hospital- Meyerstein Institute, London, England, United Kingdom

REFERENCES:
- [Result] Harland SJ: A randomised trial of radical radiotherapy in pT1G3 NXM0 bladder cancer (MRC BS06). [Abstract] J Clin Oncol 23 (Suppl 16): A-4505, 379s, 2005.